CLINICAL TRIAL: NCT01426685
Title: Prediction of Cardiovascular Events in Type 2 Diabetic Patients With Coronary Artery Disease- Application of Novel Risk Markers and Technology
Brief Title: Prognosis of Type 2 Diabetic Patients
Acronym: ARTEMIS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oulu (Other)
Collaborators: The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1539/31/06; 40042/07 (Other: Finnish Funding Agency for Technology and Innovation)
Record Dates: First submitted 2011-08-16; First posted 2011-08-31 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Risk Assessment
Keywords: sudden death; coronary artery disease; diabetes
MeSH Terms: conditions — Death, Sudden; Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are stored for analysis of various biomarkers and for extracting DNAs.
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will include 1200 patients with type 2 diabetes and angiographically documented coronary artery disease and 600 matched non-diabetic patients without type 2 diabetes. Extensive traditional and novel risk marker tests are performed for the patients and they will be followed-up for 5 years. Sudden cardiac death is the main outcome measure and various other endpoints are secondary endpoints. As a substudy, 120 diabetic patients and 120 non-diabetic patients will undergo exercise training with home monitoring to assess the effects of exercise training on risk profiles.

DETAILED DESCRIPTION:
Specific aims of the study:

1. To compare several autonomic, electric and metabolic risk markers in a case-control study between the patients with coronary artery disease with and without type II diabetes at the time of diagnosis of CAD.
2. To assess the prognostic significance of autonomic markers, electrical markers, coronary angiographic markers and metabolic markers in predicting the cardiac events among the CAD patients with and without diabetes
3. To develop and test the feasibility of home-monitoring of biosignals among the type II diabetic patients with CAD.
4. To further explore the molecular, cellular and genetic factors that predispose diabetics to cardiovascular diseases.
5. To develop new methods for the early clinical diagnosis of vulnerable subjects susceptible to the complications of the coronary artery disease in Type 2 diabetes.

5. To assess the effects of controlled exercise training programs to several autonomic, electrical and metabolic risk markers among the type II diabetic patients with CAD

ELIGIBILITY:
Inclusion Criteria:

* A total of 1200 patients with CAD and diagnosed type II diabetes and 600 patients with CAD but without evidence of diabetes will be included in the study. The patients will be recruited from the consecutive series of patients undergoing coronary angiography in the division of cardiology of the Oulu University Hospital. First, 600 patients with diabetes will be collected. Thereafter, 600 matched CAD patients without diabetes will be recruited. The groups will be matched in terms of following variables:

  1. sex (1:1)
  2. age (<40 years, 40-50 years, 50-60 years, 60-70 years, 70-80 years)
  3. history of recent (<3 months) myocardial infarction (1:1)
  4. type of coronary intervention after angiography (1:1 CABG ).
* Diabetes is defined as fasting plasma glucose levels ≥ 7.0 and/or a 2-h postload value in the OGTT 11.1 mmol/l according to definition and diagnosis of diabetes mellitus and intermediate hyperglycemia : report of a WHO/IDF consultation. World Health Organization (WHO) 2006. -
* Patients without a diabetes must be normoglycemic defined as plasma glucose levels <6.1 mmol/l in the fasting state and a 2-h postload value < 7.8 mmol/l in the oral glucose tolerance test (OGTT).

Exclusion Criteria:

* • NYHA class IV despite appropriate treatment of heart failure;

  * Planned ICD implantation;
  * Participation in a competing clinical trial that is not accepted by the Steering Committee;
  * Psychologically or physically (due to any other illness) unfit for participation in the study according to the opinion of the investigator;
  * Patient compliance doubtful;
  * Patients who are geographically or otherwise inaccessible for follow-up;
  * Pregnancy;
  * Life expectancy < 1 year;
  * end-stage renal failure needing dialysis
  * age < 18 years, or > 80 years
  * permanent pacemaker or implantable cardioverter-defibrillator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1200 diabetic patients with coronary artery disease and 600 non-diabetic patients with coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 1880 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
sudden cardiac death | 2007-2017 (up to ten years)
  Death occuurring within one hour after onset of symptoms, or within 24 hours when the patient has last seen alive

SECONDARY OUTCOMES:
cardiovascular mortality | 2007-2017 (up to ten years)
  Sudden and non-sudden cardiac death, stroke mortality
non-fatal cardiovascular event | 2007-2017 (up to ten years)
  acute coronary event, myocardial infarction, congestive heart failure, or stroke needing hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Heikki V Huikuri, MD, Principal Investigator — University of Oulu
Locations (1):
- University of Oulu, Oulu, Finland

REFERENCES:
- [Derived] Rahunen R, Tulppo M, Rinne V, Lepojarvi S, Perkiomaki JS, Huikuri HV, Ukkola O, Junttila J, Hukkanen J. Liver X Receptor Agonist 4beta-Hydroxycholesterol as a Prognostic Factor in Coronary Artery Disease. J Am Heart Assoc. 2024 Mar 5;13(5):e031824. doi: 10.1161/JAHA.123.031824. Epub 2024 Feb 23. PMID 38390795
- [Derived] Tulppo MP, Kiviniemi AM, Lahtinen M, Ukkola O, Toukola T, Perkiomaki J, Junttila MJ, Huikuri HV. Physical Activity and the Risk for Sudden Cardiac Death in Patients With Coronary Artery Disease. Circ Arrhythm Electrophysiol. 2020 Jun;13(6):e007908. doi: 10.1161/CIRCEP.119.007908. Epub 2020 May 20. PMID 32433894
- [Derived] Kiviniemi AM, Tulppo MP, Junttila MJ, Huikuri HV. Response to Comment on Kiviniemi et al. Prediabetes and Risk for Cardiac Death Among Patients With Coronary Artery Disease: The ARTEMIS Study. Diabetes Care 2019;42:1319-1325. Diabetes Care. 2019 Dec;42(12):e195. doi: 10.2337/dci19-0050. No abstract available. PMID 31748220
- [Derived] Kiviniemi AM, Lepojarvi ES, Tulppo MP, Piira OP, Kentta TV, Perkiomaki JS, Ukkola OH, Myerburg RJ, Junttila MJ, Huikuri HV. Prediabetes and Risk for Cardiac Death Among Patients With Coronary Artery Disease: The ARTEMIS Study. Diabetes Care. 2019 Jul;42(7):1319-1325. doi: 10.2337/dc18-2549. Epub 2019 May 10. PMID 31076416
- [Derived] Puurunen VP, Lepojarvi ES, Piira OP, Hedberg P, Junttila MJ, Ukkola O, Huikuri HV. High plasma leptin levels are associated with impaired diastolic function in patients with coronary artery disease. Peptides. 2016 Oct;84:17-21. doi: 10.1016/j.peptides.2016.08.002. Epub 2016 Aug 11. PMID 27524739
- [Derived] Lepojarvi ES, Piira OP, Kiviniemi AM, Miettinen JA, Kentta T, Ukkola O, Tulppo MP, Huikuri HV, Junttila MJ. Usefulness of Highly Sensitive Troponin as a Predictor of Short-Term Outcome in Patients With Diabetes Mellitus and Stable Coronary Artery Disease (from the ARTEMIS Study). Am J Cardiol. 2016 Feb 15;117(4):515-521. doi: 10.1016/j.amjcard.2015.11.038. Epub 2015 Dec 6. PMID 26739392
- [Derived] Kiviniemi AM, Lepojarvi S, Kentta TV, Junttila MJ, Perkiomaki JS, Piira OP, Ukkola O, Hautala AJ, Tulppo MP, Huikuri HV. Exercise capacity and heart rate responses to exercise as predictors of short-term outcome among patients with stable coronary artery disease. Am J Cardiol. 2015 Nov 15;116(10):1495-501. doi: 10.1016/j.amjcard.2015.08.014. Epub 2015 Aug 31. PMID 26381535
- [Derived] Karjalainen JJ, Kiviniemi AM, Hautala AJ, Piira OP, Lepojarvi ES, Perkiomaki JS, Junttila MJ, Huikuri HV, Tulppo MP. Effects of physical activity and exercise training on cardiovascular risk in coronary artery disease patients with and without type 2 diabetes. Diabetes Care. 2015 Apr;38(4):706-15. doi: 10.2337/dc14-2216. Epub 2015 Jan 15. PMID 25592198
- [Derived] Perkiomaki J, Exner DV, Piira OP, Kavanagh K, Lepojarvi S, Talajic M, Karvonen J, Philippon F, Junttila J, Coutu B, Huikuri H. Heart Rate Turbulence and T-Wave Alternans in Patients with Coronary Artery Disease: The Influence of Diabetes. Ann Noninvasive Electrocardiol. 2015 Sep;20(5):481-7. doi: 10.1111/anec.12244. Epub 2015 Jan 15. PMID 25589197